CLINICAL TRIAL: NCT07207044
Title: FAXAGE: A Randomized, Controlled Clinical Trial Of Fasting And Exercise To Slow Aging In Humans
Brief Title: FAXAGE: Fasting And Exercise To Slow Aging In Humans
Acronym: FAXAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-25020642
Record Dates: First submitted 2025-09-23; First posted 2025-10-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Aging; Healthy Aging; Aging Frailty
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TRF (Experimental)
  Interventions: Behavioral: Time-restricted feeding
- EXE (Experimental)
  Interventions: Behavioral: Exercise - Strength + Cardio
- FAX (Experimental)
  Interventions: Behavioral: Time-restricted feeding + Exercise
- CON (No Intervention)

INTERVENTIONS:
Behavioral: Exercise - Strength + Cardio — Supervised strength training 2x/week + self-administered cardio training 2x/week.
  Arms: EXE
Behavioral: Time-restricted feeding — Time-restricted feeding in a 16/8 regimen - 16 hours of fast and 8 hours of eating per day.
  Arms: TRF
Behavioral: Time-restricted feeding + Exercise — Strength and cardio exercise 2x/week each combined with time-restricted feeding in a 16/8 regimen.
  Arms: FAX

SUMMARY:
FAXAge is a randomized controlled trial investigating the effects of fasting and exercise on human aging. 240 participants over the age of 65 will be divided into 4 groups - an exercise group, a fasting group, a combined exercise and fasting group and a control group. The intervention will last for one year, and tests of biomarkers of aging will be performed at baseline, after 3 months, 6 months and at the end of the intervention. A reference group of participants over the age of 20 equally distributed by age and sex will be used to train an algorithm for determination of biological age. The study will include both physical, molecular and digital biomarkers including DNA-methylation, VO2max, body composition and face- and voice-age. The main outcome of the project is DNA-methylation age at week 52. Secondary outcomes are the rest of the tested biomarkers at week 52. It is hypothesised that the intervention groups will have similar superior benefits after the 52 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged >20 years
* In good general health meaning maximally 1 well-managed chronic disease
* Non-smoker.

Exclusion Criteria:

* Inability or unwillingness to adhere to the TRF regiment
* Inability or unwillingness to perform the prescribed physical exercise
* Treatment with other investigational drug or intervention within 1 year
* >1 hour of systematic strenuous exercise or strength training a week
* Current time-restricted eating habits
* Severe or dysregulated medical disease (i.e. active cancer, uncontrolled diabetes, severe pulmonary or heart disease)
* >1 well-managed chronic disease
* Smoker
* Use of systemic glucocorticoids, androgens or antiandrogens.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2042-08-30 (Estimated)

PRIMARY OUTCOMES:
DNA-methylation age | From enrollment until end of intervention at 52 weeks
  Changes in predicted biological age from baseline based on DNA-methylation from isolated peripheral blood mononucleated cells after 52 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Copenhagen N, Denmark